CLINICAL TRIAL: NCT05973773
Title: Randomized, Controlled, Open-label, Phase 3, Global Multi - Center Trial to Assess the Efficacy and Safety of Zipalertinib Plus Chemotherapy Versus Chemotherapy Alone, in Patients With Previously Untreated, Locally Advanced or Metastatic Nonsquamous Non-Small Cell Lung Cancer (NSCLC) With Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertion (ex20ins) Mutations
Brief Title: REZILIENT3 (REsearching ZIpaLertinib In Egfr Non-small Cell Lung Cancer Tumors)
Acronym: REZILIENT3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAS6417-301; 2023-503575-21 (EudraCT Number)
Record Dates: First submitted 2023-07-11; First posted 2023-08-03 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Advanced or Metastatic NSCLS With Exon 20 Insertion Mutation
Keywords: Exon 20 insertion mutation; NSCLC; phase 3; Lung disease; Carcinoma, Non-Small-Cell Lung; CLN-081; TAS6417; EGFR
MeSH Terms: conditions — Lung Diseases; Carcinoma, Non-Small-Cell Lung | interventions — zipalertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A (Safety Lead in) (Experimental): Part A: Safety Lead-In Approximately 6-12 patients will receive zipalertinib administered at an initial dose of zipalertinib PO BID (Dose Level 1) in combination with pemetrexed and carboplatin or cisplatin on a 21-day cycle. Patients may continue to receive study treatment until documentation of progressive disease (PD) or until other withdrawal criteria are met, whichever comes first.
  Interventions: Drug: TAS6417
- Part B (Experimental): Enrollment into the Phase 3 portion of the study will begin following completion of Part A.
  Approximately 260 patients will be randomized on a 1:1 basis to receive pemetrexed and a platinum agent (either carboplatin or cisplatin) with or without zipalertinib on a 21-day cycle.
  Carboplatin or cisplatin will be administered for 4 cycles. Patients may continue to receive zipalertinib (experimental study arm) and pemetrexed (both study arms) until documentation of PD or until other withdrawal criteria are met, whichever comes first.
  Interventions: Drug: TAS6417

INTERVENTIONS:
Drug: TAS6417 — oral tablets
  Other Names: Zipalertinib; CLN-081

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of zipalertinib in combination with standard first-line platinum-based chemotherapy compared to chemotherapy alone, in patients with locally advanced or metastatic NSCLC with EGFR ex20ins mutations.

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of zipalertinib in combination with standard chemotherapy with pemetrexed and a platinum agent (either carboplatin or cisplatin) in patients with previously untreated, locally advanced or metastatic nonsquamous NSCLC harboring EGFR ex20ins mutations.

The study will be conducted in two parts:

* Part A: Safety lead-in to determine the recommended dose of zipalertinib in combination with standard chemotherapy pemetrexed and a platinum agent (either carboplatin or cisplatin) to be studied in Part B of the study.
* Part B: Randomized, controlled, open-label, multinational Phase 3 study to assess the efficacy and safety of zipalertinib in combination with standard chemotherapy with pemetrexed and a platinum agent (either carboplatin or cisplatin) compared to standard chemotherapy alone. Patients randomized to the chemotherapy-only treatment arm in Part B may receive treatment with zipalertinib as monotherapy after BICR-assessed progressive disease (PD) is documented (optional "crossover arm").

An independent data monitoring committee (IDMC) will be established to monitor interim safety Data.

A treatment cycle is defined as 21 days for both parts of the study.

Part A: Safety Lead-In The primary objective of Part A is to determine the recommended dose of zipalertinib administered in combination with pemetrexed and a platinum agent (either carboplatin or cisplatin) to be studied in the Phase 3 portion of this study.

Approximately 6-12 patients will receive zipalertinib administered at an initial dose of zipalertinib PO BID (Dose Level 1) in combination with pemetrexed and carboplatin or cisplatin on a 21-day cycle. Patients may continue to receive study treatment until documentation of progressive disease (PD) or until other withdrawal criteria are met, whichever comes first. Patients will be enrolled using a rolling-6 design,35 and the determination of the dose of zipalertinib to be used in Part B of the study will be informed by the incidence of dose-limiting toxicities (DLTs) observed during Cycle 1.

Part B: Phase 3 Enrollment into the Phase 3 portion of the study will begin following completion of Part A.

Approximately 260 patients will be randomized on a 1:1 basis to receive pemetrexed and a platinum agent (either carboplatin or cisplatin) with or without zipalertinib on a 21-day cycle.

Carboplatin or cisplatin will be administered for 4 cycles. Patients may continue to receive zipalertinib (experimental study arm) and pemetrexed (both study arms) until documentation of PD or until other withdrawal criteria are met, whichever comes first.

ELIGIBILITY:
Inclusion-

1. Provide written informed consent.
2. ≥18 years of age (or meets the country's regulatory definition for legal adult age, whichever is greater).
3. Pathologically confirmed, locally advanced or metastatic nonsquamous NSCLC
4. Has not received any prior systemic treatment for their locally advanced or metastatic nonsquamous NSCLC. Prior adjuvant/neoadjuvant treatment received >6 months prior to first dose of study treatment is allowed for early-stage

   NSCLC. Prior monotherapy with an approved EGFR TKI (ie, gefitinib, erlotinib, afatinib, dacomitinib, or osimertinib) as nonstandard first-line therapy for the treatment of locally advanced or metastatic disease is allowed if all of the following criteria are met:
   1. Treatment duration did not exceed 8 weeks;
   2. Lack of disease response was documented (radiographically) by an increase in tumor burden (a copy of the computerized tomography [CT] report showing increase in tumor burden from baseline should be submitted);
   3. Associated toxicities have resolved to baseline; and
   4. The EGFR TKI was discontinued at least 2 weeks or 4 half-lives prior to randomization, whichever is longer.

   Prior therapy with EGFR TKI agents targeting exon20ins mutations including amivantamab, mobocertinib, sunvozertinib, furmonertinib, and poziotinib is not allowed.
5. Documented EGFR mutation status, as determined by local testing performed at a CLIA certified (US) or accredited (outside of the US) local laboratory, defined as follows:

   1. Part A: EGFR ex20ins or other uncommon single or compound EGFR mutation
   2. Part B: EGFR ex20ins mutation
6. Archival tumor tissue available for submission, with minimum quantity sufficient to evaluate EGFR mutation status and, where possible, other biomarkers. Patients with insufficient tissue (details provided in laboratory manual) may be eligible following discussion with the sponsor; a fresh biopsy will not be required.
7. Patients with brain metastasis(es) who have previously received definitive local treatment and have stable central nervous system (CNS) disease (defined as being neurologically stable and off corticosteroid for at least 2 weeks prior to enrollment) are eligible. If brain metastases are diagnosed on screening imaging, the patient may be rescreened for eligibility after definitive treatment.

   b. Asymptomatic brain metastases ≤2 cm in size can be eligible for inclusion if, in the opinion of the Investigator, immediate definitive treatment is not indicated.
8. At least one measurable lesion as determined per RECIST 1.1 for patients enrolling to Part B. Patients enrolling to Part A may be enrolled without measurable disease.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
10. Adequate organ function, as defined by the laboratory value
11. Have a life expectancy of at least 3 months as assessed by the investigator.
12. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test prior to administration of the first dose of study treatment. Female patients are not considered to be of childbearing potential if they are postmenopausal (no menses for 12 months without an alternative medical cause) or permanently sterile (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).
13. Both males and females of reproductive potential must agree to use effective birth control during the study prior to the first dose and for 6 months after the last dose of study treatment or longer, based on local requirements.

Exclusion -

1. Is currently receiving an investigational drug in a clinical trial or participating in any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Prior treatment with any of the following within the specific time frame specified:

   1. Zipalertinib (TAS6417/CLN-081) at any time.
   2. Thoracic radiotherapy ≤28 days, palliative radiation of nonthoracic disease ≤14 days, or palliative radiation of a single lesion ≤7 days prior to first dose of study treatment.
   3. Major surgery (excluding placement of vascular access) ≤28 days prior to first dose of study treatment.
   4. All prescribed medication, over-the-counter medication, vitamin preparations and other food supplements, or herbal medications that are strong or moderate CYP3A4 inducers or inhibitors within 7 days prior to first dose.
3. Have any unresolved toxicity of Grade ≥2 from previous anticancer treatment in the neoadjuvant or adjuvant setting, except for Grade 2 alopecia or skin pigmentation. Patients with other chronic but stable Grade 2 toxicities may be allowed to enroll after agreement between the investigator and Sponsor.
4. Past medical history of interstitial lung disease, treatment-related pneumonitis (any grade), or any evidence of clinically active interstitial lung disease.
5. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

   1. History of congestive heart failure (CHF) Class III/IV according to the New York Heart Association (NYHA) Functional Classification .
   2. Serious cardiac arrhythmias requiring treatment.
   3. Resting corrected QT interval (QTc) >470 msec calculated using Fridericia's formula (QTcF).
6. Unable to swallow tablets or has any disease or condition that may significantly affect gastrointestinal (GI) absorption of zipalertinib (such as inflammatory bowel disease, malabsorption syndrome, or prior GI resection).
7. History of another primary malignancy ≤2 years prior to the date of first dose of study treatment unless at least one of the following criteria are met:

   1. Adequately treated basal or squamous cell carcinoma of the skin
   2. Cancer of the breast or cervix in situ
   3. Previously treated malignancy, if all treatment for that malignancy was completed at least 2 years prior to first dose of study treatment, and no current evidence of disease
   4. Concurrent malignancy determined to be clinically stable and not requiring tumor directed treatment
8. Known history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) that is unstable or not controlled with treatment.
9. History of COVID-19 infection within 4 weeks prior to enrolment and/or have persistent, clinically significant pulmonary symptoms related to prior COVID-19 infection.
10. Active bleeding disorders.
11. Known hypersensitivity to the ingredients in zipalertinib or any drugs similar in structure or class. To platinum-containing drugs (ie, cisplatin, carboplatin), pemetrexed, or any known excipients of these drugs. b. Contraindications toning drugs (ie, cisplatin, carboplatin) or pemetrexed according to the respective local labels.
12. History of leptomeningeal disease and spinal cord compression.
13. Is unable or unwilling to take dexamethasone, folic acid, and/or vitamin B12 supplementation during treatment with pemetrexed.
14. Is pregnant or lactating or planning to become pregnant
15. The patient is, in the investigator's opinion, unable or unwilling to comply with the trial procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-10-29 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
Part A and B: The rate and severity of treatment emergent AEs | approximately 5 years
Part A and Part B: Progression-free survival (PFS) by blinded independent central review (BICR) | approximately 5 years
Part A: The rate and severity of DLTs according to the NCI-Common Terminology Criteria of Adverse Events (CTCAE) v5.0 during Cycle 1 | approximately 5 years

SECONDARY OUTCOMES:
Part A and Part B: Objective response rate (ORR) | approximately 5 years
Part A and Part B: Disease control rate (DCR) | approximately 5 years
Part A and Part B: Duration of response (DoR) | approximately 5 years
Part A and Part B: Intracranial (i) Overall Response Rate (iORR) | approximately 5 years
Part A and Part B: Intracranial duration of complete response (iDCR) | approximately 5 years
Part A and Part B: Intracranial duration of Response (iDoR) | approximately 5 years
Part B: Overall survival (OS) | approximately 5 years
Pharmacokinetic (PK) parameter | approximately 5 years
  Minimum observed concentration (Cmin)
European Quality of Life 5 Dimensions, 3 Level Version (EQ-5D-3L) | approximately 5 years
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. This scale is numbered from 0 to 100. The higher the score the better the outcome
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30 | approximately 5 years
  The EORTC QLQ-C30 is a "core questionnaire" which incorporates a range of physical, emotional and social health developed to assess the quality of life of cancer patients. This scale is numbered from 30 to 130. The higher the score equates to better functioning.
Non-small Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ ) | approximately 5 years
  The NSCLC- SAQ was developed to incorporate the patient's perspective into evaluation of clinical benefit in advanced non-small cell lung cancer trials.. Qualitative evidence supports 7 items covering 5 symptom concepts with the total score measuring overall severity of the following NSCLC symptoms: cough, pain, dyspnea, fatigue, and appetite. Lower scores indicate lower symptom severity.

OTHER OUTCOMES:
Pharmacokinetic (PK) parameter | approximately 5 years
  Minimum Plasma Concentration [Cmin]
Pharmacokinetic (PK) parameter | approximately 5 years
  Maximum Plasma Concentration [Cmax]
Pharmacokinetic (PK) parameter | approximately 5 years
  Area Under Curve [AUC]
EGFR mutation status | approximately 5 years
  local central tests results

CONTACTS AND LOCATIONS:
Locations (131):
- United States (10):
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Horizon Ridge Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Southeast Henderson - Stephanie, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Summerlin Medical Center II, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Southwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley - Twain, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Gabrail Cancer and Research Center, Canton, Ohio
  - The Toledo Clinic Cancer Center, Toledo, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (4):
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Flemish Brabant
  - Algemeen Ziekenhuis Maria Middelares, Ghent, Oost-Vlaaderen
  - Algemeen Ziekenhuis Delta - Campus Menen, Menen, West Flanders
  - Algemeen Ziekenhuis Delta - Campus Rumbeke, Rosières, West-Vlaanderen
- Brazil (5):
  - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Hospital Mãe de Deus - Centro Integrado de Oncologia, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Clínica Neoplasias Litoral, Itajaí, Santa Catatina
  - Hospital Amaral Carvalho, Jaú, São Paulo
- Bulgaria (2):
  - Multi-profile Hospital for Active Treatment Uni Hospital, Panagyurishte, Pazardzhik
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna-ISUL, Sofia
- Canada (3):
  - BC Cancer Vancouver, Vancouver, British Columbia
  - William Osler Health System - Brampton Civic Hospital, Brampton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Chile (3):
  - CentroEstudiosClinicosSAGA, Santiago, Region de Santiago
  - Hospital Clínico Universidad de Chile, Independencia, Santiago Metropolitan
  - Instituto Oncológico Fundación Arturo López Pérez, Providencia, Santiago Metropolitan
- France (9):
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace
  - Hôpital Côte De Nacre, Caen, Basse-Normandie
  - Centre Hospitalier Universitaire Limoges, Limoges, Limousin
  - Hôpital Haut-Lévêque, Pessac, Nouvelle-Aquitaine
  - Centre Hospitalier Le Mans, Le Mans, Pays de la Loire Region
  - Gustave Roussy, Villejuif, Val-de-Marne
  - CH Cornouaille Quimper, Quimper
  - Hôpital Ambroise-Paré, Boulogne-Billancourt, Île-de-France Region
  - Institut Curie, Paris, Île-de-France Region
- Germany (4):
  - Asklepios Klinik Altona, Hamburg, Hamburg (Hansestadt)
  - Universitätsklinikum Gießen und Marburg - Gießen, Giessen, Hesse
  - LMU Klinikum - Campus Innenstadt, München
  - Universitätsklinikum Regensburg, Regensburg
- Greece (6):
  - General Hospital for Thoracic Diseases Sotiria, Athens, Attica
  - Metropolitan General, Piraeus, Attica
  - University General Hospital of Patras, Patra, Peloponnese
  - Metropolitan Hospital, Piraeus, Pireas
  - University General Hospital of Larissa, Larissa, Thessaly
  - BioClinic Thessaloniki, Thessaloniki
- Israel (5):
  - Emek Medical Center, Afula
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Hospital - Ramat HaHayal, Tel Aviv
- Italy (9):
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST, Meldola, Forli-Cesena
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST, Meldola, Forlì-Cesena
  - Istituto Nazionale per la Ricerca sul Cancro, Genova, Genoa
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero - Universitaria di Modena, Modena
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Unità Sanitaria Locale della Romagna, Ravenna
  - IRCCS Istituto Nazionale Tumori Regina Elena, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (15):
  - Aichi Cancer Center, Nagoya, Aiti [Aichi]
  - Hirosaki University Hospital, Hirosaki-Shi, Aomori
  - Kyushu Cancer Center, Fukuoka, Hukuoka
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai-Shi, Osaka
  - Cancer Institute Hospital of JFCR, Koto, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Kanazawa University Hospital, Kanazawa
  - Osaka City General Hospital, Osaka
  - Osaka Prefectural Hospital Organization - Osaka International Cancer Institute, Osaka
- Mexico (6):
  - Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco
  - Actualidad Basada en la Investigación del Cáncer, Guadalajara, Jalisco
  - Health Pharma Professional Research S.A. De C.V, Mexico City, Mexico City
  - Clínica Integral Internacional de Oncología S de RL de CV, Mirador, Puebla
  - Investigacion Medica Galerias, Aguascalientes
  - FAICIC Clínical Research, Veracruz
- Netherlands (3):
  - Radboud Universitair Medisch Centrum, Nijmegen, Gelderland
  - Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, North Holland
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
- Philippines (3):
  - St. Luke's Medical Center - Quezon City, Quezon City, Metropolitan Manila
  - The Medical City, Pasig, National Capital Region
  - Asian Hospital and Medical Center, City of Muntinlupa
- Poland (3):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im. Eugenii i Janusza Zeylandów, Pozna?, Greater Poland Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin, Lublin Voivodeship
  - Instytut MSF, Lodz, Lódzkie
- Romania (4):
  - Medisprof, Cluj-Napoca, Cluj
  - Centrul de Oncologie Sf Nectarie, Craiova, Dolj
  - Oncocenter - Oncologie Clinica, Timișoara, Timiș County
  - Clinica SIGMedical, Suceava
- Singapore (5):
  - National Cancer Centre Singapore, Singapore
  - Icon Cancer Centre - Mount Alvernia, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Oncocare Cancer Centre, Singapore
  - Icon Cancer Centre Mount Elizabeth, Singapore
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Catholic University of Korea Saint Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnamdo [Kyongsangnam-do]
  - Inha University Hospital, Incheon, Incheon Gwang'yeogsi [Inch'on-Kwangyokshi]
  - Korea University Anam Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
- Spain (10):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Clínica Mi Tres Torres, Barcelona
  - Hospital Quirónsalud Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Jaén, Jaén
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga - Hospital General, Málaga
- Thailand (3):
  - Faculty of Medicine Siriraj Hospital, Bang Phlat, Bangkok
  - King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok
  - Navamindradhiraj University - Faculty of Medicine Vajira Hospital, Bangkok, Khet Dusit
- Turkey (Türkiye) (9):
  - T.C. Saglik Bakanligi Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Medical Park Seyhan Hastanesi, Adana
  - Hacettepe Üniversitesi Kanser Enstitüsü, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - T.C. Saglik Bakanligi Ankara Bilkent Sehi?r Hastanesi?, Çankaya
  - Trakya Üniversitesi Sa?l?k Ara?t?rma ve Uygulama Merkezi, Edirne
  - Ankara Il Saglik Mudurlugu SBU Gulhane Egitim Ve Arastirma Hastanesi, Etlik
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - T.C. Saglik Bakanligi - Istanbul Il Saglik Mudurlugu - Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
- United Kingdom (3):
  - Royal Free London NHS Foundation Trust, London, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England
  - Torbay and South Devon NHS Foundation Trust, Torquay, England

REFERENCES:
- [Derived] Heymach JV, Yu HA, Besse B, Cheng Y, Tan DS, Wei L, Wacheck V, Nishio M. REZILIENT3: randomized phase III study of first-line zipalertinib plus chemotherapy in patients with EGFR exon 20 insertion-mutated NSCLC. Future Oncol. 2025 Feb;21(5):549-556. doi: 10.1080/14796694.2025.2457294. Epub 2025 Feb 16. PMID 39957151